CLINICAL TRIAL: NCT07270198
Title: Longitudinal Multicentre Clinical Study to Explore the Mechanisms Underlying Kidney Effect of SGLT2i in Diabetic Kidney Disease Patients at Risk of Disease Progression by Multiparametric Renal MRI and Biochemical Markers
Brief Title: Mechanisms Underlying SGLT2i Kidney Effect in DKD Progression
Acronym: PERSONALISEDKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PERSONALISE-DKD
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Kidney Disease (DKD)
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Adult Diabetic Kidney Disease (DKD) patients with CKD stages 1 to 3 at moderate or severe risk of renal disease progression.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Multiparametric non-contrast enhanced renal MRI and biochemical analysis to investigate MMP-related pathways (MMP-10 and TIMP-1 serum levels)

SUMMARY:
This is a multicentre and multi-national non-pharmacological, uncontrolled interventional study conducted in a clinical practice setting in DKD patients with CKD stages 1 to 3 with moderate or severe risk of renal function decline in chronic treatment with SGLT2i.

The main aim of the study is to assess the independent role of baseline individual mpMRI markers (hemodynamic, oxygenation, microstructure, perfusion, and fat fraction) and biochemical markers of MMP-related pathways (MMP-10 and TIMP-1) in the prediction of chronic eGFR decline in the above mentioned patients who are on chronic SGLT2i therapy.

DETAILED DESCRIPTION:
Recent years have seen an exponential increase in the incidence and prevalence of chronic kidney disease (CKD). Diabetes Mellitus is the leading cause of CKD. Diabetic kidney disease (DKD) is clinically defined by the presence of reduced kidney function and/or increased albuminuria for at least three months in patients with diabetes. However, not all patients with diabetes develop DKD and not all patients with DKD follow the same trajectory. Sodium-glucose cotransporter 2 inhibitors (SGLT2i) have recently shown significant nephroprotective benefits, making them a first-line therapy in DKD. Although the mechanisms underlying SGLT2i nephroprotection are not fully understood, preliminary data suggest a long-term benefit on metabolic, haemodynamics, and/or kidney injury pathways. SGLT2i have also been shown to be nephroprotective in mouse models, attenuating renal fibrosis in diabetes. These promising results underscore the potential of SGLT2i to avert severe CKD events through early intervention, particularly in patients at higher risk of progression. However, clinical, and genetic factors may influence response to SGLT2i in patients with comorbid conditions and already receiving antidiabetic and antihypertensive drugs. Thus, with the scope to personalised medicine, it would be key to early identify DKD patients with rapid progressive decline in renal function that is associated with increased morbidity and mortality, who may benefit the most from SGLT2i therapy. To achieve this, biomarkers with heightened specificity and sensitivity to disease progression and response to treatment are urgently needed.

Renal multiparametric MRI (mpMRI) has recently shown great potential to investigate renal structure, microstructure, and function, facilitating the diagnosis and monitoring of CKD progression and response to treatment. Recent studies showed the ability of decreased renal blood flow - assessed by arterial spin labelling (ASL) MRI sequence - in detecting subclinical renal involvement in patients with type 2 diabetes.

Blood oxygenation level dependent (BOLD)-MRI sequence showed an acute effect on renal cortical oxygenation in response to SGLT2i treatment in type I diabetic patients with albuminuria.

mpMRI shows potential to investigate and quantify renal and perirenal adipose tissue (fat fraction), that is thought to play a significant role on the renal involvement in diabetes and obesity. mpMRI has also shown its ability to monitor the effects of SGLT2i treatment in patients with type 2 diabetes mellitus.

Moreover, the hallmark of DKD pathogenesis is increased extracellular matrix (ECM) accumulation causing thickening of the glomerular and tubular basement membranes, followed by mesangial expansion, sclerosis, and tubulointerstitial fibrosis. Dysregulated balance between levels of matrix metalloproteases (MMPs, involved in ECM degradation and hydrolysis) and their tissue inhibitors (TIMP) has been found in DKD patients, and altered serum and urine TIMP-1 levels have been linked with worsening glomerular lesions. MMP-10 null diabetic mice presented fewer mesangial expansion, renal macrophage infiltration and renal function impairment. These findings may support a deleterious kidney effect of MMP-10 in DKD.

To build on and validate these single-centre findings, a more precise risk stratification and an in-depth study of the underlying mechanisms are essential to personalise DKD renal management.

The PERSONALISE-DKD clinical study will aim at identifying and characterising DKD patients with moderate and severe risk of renal disease progression despite SGLT2i treatment, who could benefit the most from future clinical trials and health policies, possibly changing the paradigm of a disease that so far has been the main cause of advanced CKD.

ELIGIBILITY:
Inclusion Criteria (to be eligible to participate in this trial, an individual must meet all the following criteria):

* male and female subjects aged ≥ 18 years;
* written informed consent prior to any study specific procedures
* type 2 Diabetes Mellitus with DKD
* CKD stage 1 to 3 (eGFR>30 ml/min) with moderate or severe risk of renal disease progression (according to KDIGO 2024 CKD guidelines, G1 and G2 with albuminuria >300 mg/g, G3a with albuminuria >30 mg/g, and G3b independently of albuminuria levels)
* ongoing SGLT2i treatment (e.g. canagliflozin, empagliflozin or dapagliflozin) for at least 1 year and stable RAS inhibitor therapy with ACE inhibitors and/or ARBs (or without RAS inhibitors in patients with specific contraindications for this medication)

Exclusion Criteria (an individual who meets any of the following criteria will be excluded from participation in this trial):

* Uncontrolled diabetes (glycated hemoglobin (A1C) > 8%; 64 mmol/mol)
* Contraindications to MRI including claustrophobia, pregnancy or lactating, cardiac pacemakers, or other MRI-incompatible prostheses, or impossibility to perform MRI
* Any chronic clinical condition (e.g. history of malignancy) other than CKD and related complications that could affect completion of the trial or confound data interpretation
* Non-diabetic CKD: CKD highly suspected to be related with a different renal condition other than Diabetes Mellitus as the cause of CKD (i.e. glomerular disease, tubulo-interstitial nephritis, microangiopathic thrombotic disease, renovascular/ischemic kidney disease, etc)
* Active systemic autoimmune diseases
* Concomitant treatment with steroids or any other immunosuppressive agent
* Chronic heart failure with New York Heart Association class III-IV at the screening visit
* Intention to become pregnant in the following 2 years (female patients)
* Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | At day 0, at 1 month and at 18 months
  EGFR estimation by CKD-EPI and EKFC equations (ml/min)
Matrix metalloproteases (MMPs) and their tissue inhibitors (TIMP) | At day 0, at 1 month and at 18 months
  Serum levels of MMP-10 and TIMP-1 will be assessed in blood samples by commercial ELISA kits, according to the manufacturer's instructions (pg/ml)
Multiparametric kidney MRI | At day 0, at 1 month and at 18 months
  Total kidney, cortical and medullary volumes (in mL)
Multiparametric kidney MRI | At day 0, at 1 month and at 18 months
  Renal tissue oxygenation obtained by measuring the R2* relaxation rate (in 1/ms)
Multiparametric kidney MRI | At day 0, at 1 month and at 18 months
  Apparent diffusion coefficient (in cm2/s)
Multiparametric kidney MRI | At day 0, at 1 month and at 18 months
  Renal tissue perfusion (in mL/100mL/min)
Multiparametric kidney MRI | At day 0, at 1 month and at 18 months
  Renal blood flow (in mL/min)
Multiparametric kidney MRI | At day 0, at 1 month and at 18 months
  T1 and T2 relaxation times (in ms)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, M.D., Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Clinical Research Centre for Rare Diseases Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No